CLINICAL TRIAL: NCT03182374
Title: A Two-Phase, Multicenter, Randomized Study Comparing Autologous Protein Solution With Hyaluronic Acid Intra Articular Injections in Patients With Knee Osteoarthritis
Brief Title: nSTRIDE APS Versus Hyaluronic Acid for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APSS-66-00
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Autologous Protein Solution (APS); Intra-articular Injection; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: During the long-term follow-up phase (12 - 48 months), subjects may also elect to cross over to the other treatment arm and receive additional injections of the other treatment as frequently as needed, provided they did not experience any significant clinical concerns after previous treatment administrations and are benefiting from it, as determined by the investigator. Subjects may only cross over from their originally assigned treatment group to the other treatment group one time during the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study where subjects and evaluators are blinded to treatment up to 12-months. During the long-term follow-up phase (12 - 48 months), only subjects will be blinded to the study treatment resulting in single-blind design following 12-month follow-up time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- nSTRIDE APS (Active Comparator): The nSTRIDE APS Kit is designed to be used for the safe and rapid preparation of APS from a small sample of blood at the patient's point of care. The APS is to be injected intra-articularly for the treatment of knee osteoarthritis and associated symptoms.
  Interventions: Device: nSTRIDE APS
- Synvisc-One (Active Comparator): Synvisc-One is only intended for intra-articular use by a physician to treat pain associated with osteoarthritis of the knee
  Interventions: Device: Synvisc-One

INTERVENTIONS:
Device: nSTRIDE APS — Intra-articular injection
  Other Names: Autologous Protein Solution
  Arms: nSTRIDE APS
Device: Synvisc-One — Intra-articular injection
  Other Names: hylan G-F 20
  Arms: Synvisc-One

SUMMARY:
This is a two-phase multicenter, double-blind, randomized, prospective evaluation of intra-articular injection(s) comparing APS to intra-articular HA injection(s). The maximum study duration for each subject will be 50 months; 48 months from treatment to last follow-up, and two additional months if the maximum visit window is realized. A total of 246 patients will be enrolled. These patients will meet specific inclusion and exclusion criteria, but can be generally characterized as patients with painful unilateral knee OA who have been unable to achieve satisfactory pain relief with previous conservative OA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at time of screening.
* Willingness and ability to comply with study procedures and visit schedules and able to follow oral and written instructions.
* A standing knee radiograph showing a K-L grade of 2 to 4
* Body mass index ≤ 40 kg/m2
* A qualifying WOMAC LK 3.1 pain subscale total score
* Signed an ethics committee-reviewed and approved informed consent form.

Exclusion Criteria:

* Presence of clinically observed active infection in the index knee
* Presence of symptomatic OA in the non-study knee at screening
* Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis secondary to other inflammatory diseases; HIV, viral hepatitis; chondrocalcinosis, Paget's disease, or villonodular synovitis
* Diagnosed with leukemia, known presence of metastatic malignant cells, or ongoing or planned chemotherapeutic treatment
* Presence of venous or lymphatic stasis in the index leg
* A history of local anesthetic allergy
* Previously documented failed treatment with nSTRIDE APS or Synvisc One

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizaveta Kon, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (14):
- AZ Monica, Antwerp, Belgium
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark
- Germany (2):
  - Praxiskliniek für Unfallchirurgie und Orthopädie, Eisenach
  - KniePraxis, Straubing
- Italy (2):
  - Rizzoli Orthopedic Institute, Bologna
  - The Istituto Clinico Humanitas, Milan
- Maastricht UMC+, Maastricht, Netherlands
- Oslo University Hospital - Olympiatoppen, Oslo, Norway
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
- Ospedale Regionale di Lugano, Lugano, Switzerland
- Yildirim Beyazit University, School of Medicine, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Gloucestershire Hospitals NHS Foundation Trust, Cheltenham
  - Royal Infirmary of Edinburgh - NHS Lothian, Edinburgh

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The clinical investigation began on 25 July 2017 when the first subject received treatment. Subject recruitment was completed on 20 September 2018, when the last subject was randomized and received injection.
Pre-assignment Details: Subjects giving written informed consent underwent screening assessments including demographics, medical history, physical examination, knee examination, a urine pregnancy test (if applicable) and the WOMAC LK 3.1. Upon confirmation of eligibility, subjects were scheduled for a treatment visit, and a baseline X-ray and MRI were performed.
Groups:
- Synvisc-One: Synvisc-One is intended for intra-articular use by a physician to treat pain associated with osteoarthritis of the knee
  Synvisc-One: Intra-articular injection
Period: Overall Study
Arm/Group | nSTRIDE APS | Synvisc-One
Started | 125 | 127
Treated (Patients who received the first injection) | 124 (One subject that was randomized in the nSTRIDE group was not treated) | 127
12-month Follow-up | 111 (Fourteen (14) subjects in the nSTRIDE APS group had missing 12 Month follow-up data due to: additional invasive treatment in index knee within 12 months of initial injection (n=8), informed consent withdrawal (n=1), lost to follow-up (n=3), exit for non-compliance (n=1) and one subject was randomized but not treated (n=1)) | 106 (In the Synvisc-One group, 21 subjects had no 12 Month follow-up data due to: study exit for intolerable adverse event (AE) leading to invasive treatment in index knee (n=2), additional invasive treatment in index knee within 12 months of initial injection (n=12), informed consent withdrawal (n=1), lost to follow-up (n=2), exit for non-compliance (n=1) and study exit for other reason (n=3))
Completed (Subjects will complete after 5 years follow up) | 111 (subjects completed 12 months follow up) | 106 (subjects completed 12 months follow up)
Not Completed | 14 | 21
Not completed — Lost to Follow-up | 3 | 2
Not completed — Lack of Efficacy | 8 | 14
Not completed — Withdrawal by Subject | 1 | 1
Not completed — exit for non-compliance | 1 | 1
Not completed — one subject was randomized but not treated | 1 | 0
Not completed — Other reasons | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | nSTRIDE APS | Synvisc-One | Total
Number analyzed (Participants) | 125 | 127 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] — mean age of all enrolled subjects at time of enrollment
  years | 58.9 (10.52) | 57.9 (10.82) | 58.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 78 | 153
  Male | 50 | 49 | 99
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.20 (4.211) | 27.53 (4.217) | 27.86 (4.214)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Months Post-injection in Mean WOMAC LK3.1 Pain Score in Both Arms of the Study (nSTRIDE APS and Synvisc One)
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain (5), stiffness (2), and physical function (17). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. 0 represents the best health status and 96 the worst possible status.
  This section will only analyze the WOMAC pain score.
Time Frame: 12 months
Population: ITT population, with imputations for missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS | Synvisc-One
Number analyzed (Participants) | 125 | 127
score on a scale
  Baseline | 11.5 (2.36) | 11.9 (2.45)
  12 month Follow-up: number analyzed (Participants) | 111 | 106
  12 month Follow-up | 6.7 (3.93) | 7.2 (4.26)
Statistical Analysis 1: Comparison: nSTRIDE APS vs Synvisc-One; Test type: Superiority; p < 0.0001, t-test, 2 sided — ITT Population

2. Secondary Outcome: Change From Baseline to 12 Months Post-injection in Mean NRS Pain Scale in Both Arms of the Study (nSTRIDE APS and Synvisc One)
Description: In a Numerical Rating Scale (NRS) pain scale, patients are asked to circle (in an horizontal bar or line) the number between 0 and 10 that fits best to their average pain intensity.
  0 = No pain at all; 5 = Moderate pain; 10 = Worst possible pain
Time Frame: 12 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS | Synvisc-One
Number analyzed (Participants) | 102 | 98
score on a scale
  Baseline | 5.8 (2.0) | 6.2 (1.8)
  12 month follow-up: number analyzed (Participants) | 101 | 98
  12 month follow-up | 4.0 (2.53) | 4.4 (2.51)
Statistical Analysis 1: Comparison: nSTRIDE APS vs Synvisc-One; Test type: Superiority; p < 0.0001, t-test, 2 sided — PP Population

3. Secondary Outcome: Number or Participants Achieving Clinical Success as Defined by OMERACT-OARSI Responder Criteria in Both Arms of the Study (nSTRIDE APS and Synvisc One)
Description: The Outcome Measures in Rheumatology workgroup (OMERACT), together with the Osteoarthritis Research Society International (OARSI) developed the OMERACT-OARSI responder criteria. These criteria are used to determine if a patient with osteoarthritis (OA) 'responds' to therapy, meaning experiences a clinically relevant effect of therapy.
  It includes three symptomatic domains (pain, function, and patient's global assessment).
  To the question: High improvement in pain or in function (≥50%) and absolute change ≥20%, a positive answer is understood as "Response". A negative answer leads to an additional analysis, which seeks improvement in at least 2 of the 3 following:
  1. pain ≥20% and absolute change ≥10;
  2. function ≥20% and absolute change ≥10;
  3. patient's global assessment ≥20% and absolute change ≥10. A positive answer here is understood as "Response". A negative answer is a "No response"
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | nSTRIDE APS | Synvisc-One
Number analyzed (Participants) | 102 | 98
Participants
  Responder | 60 | 61
  Non-responder | 42 | 37
Statistical Analysis 1: Comparison: nSTRIDE APS vs Synvisc-One; Test type: Superiority; p = 0.6655, t-test, 2 sided — PP Population

4. Secondary Outcome: Change From Baseline to 12 Months Post-injection in Mean WOMAC LK 3.1 Function Subscale in Both Arms of the Study (nSTRIDE APS and Synvisc One)
Description: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain (5), stiffness (2), and physical function (17). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. The sum of the scores for all three subscales gives a total WOMAC score.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. 0 represents the best health status and 96 the worst possible status.
  This section will analyze the WOMAC Function subscale. A subject is considered an MCID Function responder if they show an absolute improvement of >= 20 points in WOMAC Function from baseline to 12 Months.
Time Frame: 12 months
Population: MCID Function Responder analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS | Synvisc-One
Number analyzed (Participants) | 102 | 98
score on a scale
  Baseline | 35.4 (11.47) | 39.5 (11.60)
  12 month follow-up | 20.5 (13.46) | 23.0 (14.62)
Statistical Analysis 1: Comparison: nSTRIDE APS vs Synvisc-One; Test type: Superiority; p < 0.0001, t-test, 2 sided — PP Population

5. Secondary Outcome: Change From Baseline to 12 Months Post-injection in Mean EQ-5D in Both Arms of the Study (nSTRIDE APS and Synvisc One) - VAS Score
Description: The EurpoQol five-dimensional (EQ-5D) is a standardized instrument for measuring the health-related quality of life.
  Part of the Eq-5Q questionnaire consist of a visual analogue score (VAS), a vertical calibrated line, on which a patient rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health). Respondents indicate where they perceive their present state of health to lie, relative to these anchors.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS | Synvisc-One
Number analyzed (Participants) | 102 | 98
score on a scale
  Baseline | 68.7 (16.92) | 68.0 (16.88)
  12 month follow-up | 73.4 (16.02) | 71.7 (16.80)
Statistical Analysis 1: Comparison: nSTRIDE APS vs Synvisc-One; Test type: Superiority; p < 0.05, t-test, 2 sided — PP population

6. Secondary Outcome: Change From Baseline to 12 Months Post-injection in Mean EQ-5D in Both Arms of the Study (nSTRIDE APS and Synvisc One) - Health Status Score
Description: The EurpoQol five-dimensional (EQ-5D), section Health Status, is a standardized instrument for measuring the health-related quality of life, which assesses health status in terms of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety depression. Each question has five levels of response (no problem, slight problem, moderate problems, severe problems, extreme problems/unable to), which are singularly rated and then combined into a health status score. The health status ranges from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher score indicating higher health utility.
Time Frame: 12 months
Population: patients lost during follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS | Synvisc-One
Number analyzed (Participants) | 102 | 98
score on a scale
  Baseline | 0.6 (0.27) | 0.6 (0.27)
  12 month follow-up: number analyzed (Participants) | 102 | 97
  12 month follow-up | 0.7 (0.20) | 0.7 (0.24)
Statistical Analysis 1: Comparison: nSTRIDE APS vs Synvisc-One; Test type: Superiority; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: During the first phase of the study (up to 12 Months), all AEs were collected regardless of relationship to the device.
Arm/Group | nSTRIDE APS | Synvisc-One
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/127
Serious Adverse Events (participants affected / at risk) | 8/124 | 9/127
Other Adverse Events (participants affected / at risk) | 34/124 | 21/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | nSTRIDE APS (N=124) | Synvisc-One (N=127)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 0 | 1
Medial Meniscus Lesion+Cartilage Lesion at Medial Femoral Condyle Left Knee (Musculoskeletal and connective tissue disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Wrist affected (Musculoskeletal and connective tissue disorders) | 1 | 0
Biceps tendon rupture right arm (Musculoskeletal and connective tissue disorders) | 0 | 1 — After accident
Accute appendicitis (Gastrointestinal disorders) | 1 | 0
Infection index knee (Musculoskeletal and connective tissue disorders) | 0 | 1
Excessive swelling of Index Knee (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercalcemia (Blood and lymphatic system disorders) | 0 | 1
Actinic and Seborhoeic Keratosis in scalp and right ear (Skin and subcutaneous tissue disorders) | 1 | 0
Hospital admission for gout in left (non index knee) (Musculoskeletal and connective tissue disorders) | 1 | 0
Worsening of arthrosis left (non index) knee (Musculoskeletal and connective tissue disorders) | 1 | 0
gyneacological operation myom ovaries benigne (Reproductive system and breast disorders) | 0 | 1
Excessive pain of index knee (Musculoskeletal and connective tissue disorders) | 0 | 1
Ureteral colic (kidney stones) (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | nSTRIDE APS (N=124) | Synvisc-One (N=127)
Injection site swelling (General disorders) | 1 | 0
Vessel puncture site bruise (General disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Injection site pain (Injury, poisoning and procedural complications) | 8 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11
Joint stiffness (Musculoskeletal and connective tissue disorders) | 4 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 10 | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Venipuncture (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT03182374/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT03182374/SAP_001.pdf